CLINICAL TRIAL: NCT01997034
Title: Physiological Factors That Influence Maintenance of Lifestyle Changes and Weight Loss - a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Ubberup Folk High School (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Ph.D., Associate Professor, University of Copenhagen
Other Study IDs: UBBERUP 3
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Overweight
Keywords: Weight loss maintenance; Body composition; Physical activity; Lifestyle intervention
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, muscle and fat tissue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intensive Lifestyle Intervention: Former participants of Ubberup Folk High Schools intensive lifestyle intervention programme.
  Interventions: Behavioral: Intensive Lifestyle Intervention

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — The included subjects has previously participated in the Intensive Lifestyle Intervention intervention at Ubberup Folk High School. This intervention includes daily exercise and a hypocaloric diet (app. -700KCal/day) for 10-14 weeks. Furthermore theoretical and practical education within e.g. Nutrition, exercise and motivational psychology.

SUMMARY:
In Denmark and the western world, there is an increasing prevalence of obesity probably due to a combination of inadequate daily physical activity and a high energy intake. One approach to achieve weight loss and change life style is to participate in an intensive supervised prolonged life style modification course. The immediate effect is often positive, but over time the overall effect is limited as the majority will not maintain weight loss and a changed life style.

The purpose of this study is therefore to characterize the physiological factors that determine/influence the capacity to maintain weight loss and a healthy lifestyle after a prolonged lifestyle intervention.

The investigators have the following research questions:

1. Are there physiological traits and characteristics that mediate better adherence to lifestyle changes and weight loss?
2. Does the adaptation in muscle oxidative capacity after lifestyle intervention predict success in maintaining weight loss and lifestyle changes?
3. How does gender and age influence the capacity to maintain the lifestyle induced adaptation in muscle and adipose tissue and maintaining weight loss?

The study design is cross-sectional and will be based on a lifestyle intervention, as it is practiced in a real life setting at Ubberup folk high school. The investigators will recruit former participants of this lifestyle style intervention. 50 % who maintained a weight loss and a healthy life style and 50 % who did not.

ELIGIBILITY:
Inclusion Criteria:

* Former participants of Ubberup Folk High School

Exclusion Criteria:

* Gastric Bypass Surgery or Gastric Banding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Former participants of Ubberup Folk High School will be included in this study. Ubberup Folk High School is a privately hold externate that teaches lifestyle intervention courses with focus on weight loss. A stay at Ubberup has a duration of 10-14 weeks and is primarily self-financed. The study population will consist of men and women of two different age Groups (18-35 and 35-65yr). We will recruit participants who succeeded in maintaining the weight loss and participants who regained in weight.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total Body weight | 0-14 years after the intervention is completed

SECONDARY OUTCOMES:
Anthropometry | 0-14 years after the intervention is completed
  Body composition measured by dual x-ray absorptiometry or bio-impedance, height, weight, waist circumference.
Maximal fat oxidation | 0-14 years after the intervention is completed
  Respiratoric Exchange Ratio (RER) is measured during an incremental cycling test and maximal fat oxidation is calculated
Maximal Oxygen Consumption | 0-14 years after the intervention is completed

OTHER OUTCOMES:
Adherence to a healthy diet | 0-14 years after the intervention is completed
  Questionnaire (24hrs dietary recall) and diary to determine adherence to a healthy diet
Adherence to physical activity | 0-14 years after the intervention is completed
  International Physical Activity Questionnaire (IPAQ) to determine adherence to physical activity. Furthermore we will use diary and ActiHeart (accelerometer).
Mitochondria respiration and efficiency | 0-14 years after the intervention is completed
  Mitochondria respiration and efficiency measured by Oreboros Oxygraph
Blood and plasma substrates, hormones and metabolites | 0-14 years after the intervention is completed
  HbA1c, insulin, leptin, glucose, adiponectin, thyroid stimulating hormone (TSH), Ghrelin.
Muscle lipid composition | 0-14 years after the intervention is completed
  Muscle lipid composition will be analyzed using a lipidomics approach.
Expression of muscle lipases | 0-14 years after the intervention is completed
  Western Blot analyses will be Applied to analyse expression of muscle lipases; hormone sensitive lipase (HSL), adipose triglyceride lipase (ATGL) and lipoprotein lipase (LPL) as well muscle PAT proteins; PLIN 2 (ADRP), PLIN 3 (TIP47) and PLIN5 (OXPAT)
Adipose tissue macrophage inflammation and cytokine production | 0-14 years after the intervention is completed
Intramuscular lipid droplet content and size, glycogen content and ceramide content and location | 0-14 years after the intervention is completed
  Intramuscular lipid droplet content and size, glycogen content and ceramide content and location wil be quantified by immunohistochemical staining of serial cryo-sections of muscle tissue samples that are visualized by confocal microscopy
Motivation for lifestyle changes and sociological factors involved | 0-14 years after the intervention is completed
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, PhD, Principal Investigator — University of Copenhagen, Department of Biomedical Sciences
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

REFERENCES:
- [Background] Karlsen TI, Sohagen M, Hjelmesaeth J. Predictors of weight loss after an intensive lifestyle intervention program in obese patients: a 1-year prospective cohort study. Health Qual Life Outcomes. 2013 Oct 3;11:165. doi: 10.1186/1477-7525-11-165. PMID 24090083
- [Background] McCormack SE, McCarthy MA, Harrington SG, Farilla L, Hrovat MI, Systrom DM, Thomas BJ, Torriani M, McInnis K, Grinspoon SK, Fleischman A. Effects of exercise and lifestyle modification on fitness, insulin resistance, skeletal muscle oxidative phosphorylation and intramyocellular lipid content in obese children and adolescents. Pediatr Obes. 2014 Aug;9(4):281-91. doi: 10.1111/j.2047-6310.2013.00180.x. Epub 2013 Jun 25. PMID 23801526
- [Background] Danielsen KK, Svendsen M, Maehlum S, Sundgot-Borgen J. Changes in body composition, cardiovascular disease risk factors, and eating behavior after an intensive lifestyle intervention with high volume of physical activity in severely obese subjects: a prospective clinical controlled trial. J Obes. 2013;2013:325464. doi: 10.1155/2013/325464. Epub 2013 Apr 22. PMID 23710347
- [Background] Bruun JM, Helge JW, Richelsen B, Stallknecht B. Diet and exercise reduce low-grade inflammation and macrophage infiltration in adipose tissue but not in skeletal muscle in severely obese subjects. Am J Physiol Endocrinol Metab. 2006 May;290(5):E961-7. doi: 10.1152/ajpendo.00506.2005. Epub 2005 Dec 13. PMID 16352667
- [Background] Pedersen JO, Zimmermann E, Stallknecht BM, Bruun JM, Kroustrup JP, Larsen JF, Helge JW. [Lifestyle intervention in the treatment of severe obesity]. Ugeskr Laeger. 2006 Jan 9;168(2):167-72. Danish. PMID 16403343
- [Background] Bruun JM, Stallknecht B, Helge JW, Richelsen B. Interleukin-18 in plasma and adipose tissue: effects of obesity, insulin resistance, and weight loss. Eur J Endocrinol. 2007 Oct;157(4):465-71. doi: 10.1530/EJE-07-0206. PMID 17893261
- [Background] Christiansen T, Bruun JM, Madsen EL, Richelsen B. Weight loss maintenance in severely obese adults after an intensive lifestyle intervention: 2- to 4-year follow-up. Obesity (Silver Spring). 2007 Feb;15(2):413-20. doi: 10.1038/oby.2007.530. PMID 17299115
- [Derived] Elsborg P, Elbe AM. Exercise-specific volition and motivation for weight loss maintenance following an intensive lifestyle intervention. Health Psychol. 2018 Aug;37(8):759-766. doi: 10.1037/hea0000636. PMID 30024231